CLINICAL TRIAL: NCT02993068
Title: Stand up to Cancer: MAGENTA (Making Genetic Testing Accessible)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual Limit
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0298; NCI-2017-01600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0298 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-02

CONDITIONS: BARD1 Gene Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; BRIP1 Gene Mutation; Estrogen Receptor Negative; HER2/Neu Negative; MLH1 Gene Mutation; MSH2 Gene Mutation; MSH6 Gene Mutation; PALB2 Gene Mutation; PMS2 Gene Mutation; Progesterone Receptor Negative; RAD51C Gene Mutation; RAD51D Gene Mutation; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (online education) (Experimental): Patients watch genetic testing online educational video and receive genetic testing online test results report.
  Interventions: Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm B (online education, post telephone counseling) (Experimental): Patients watch genetic testing online educational video, receive genetic testing online test results report, and post-telephone genetic counseling.
  Interventions: Other: Educational Intervention; Other: Genetic Counseling; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm C (online education, pre- and post-telephone counselling) (Active Comparator): Patients watch genetic testing online educational video, receive pre-telephone genetic counseling, genetic testing online test results report, and post-telephone genetic counseling.
  Interventions: Other: Educational Intervention; Other: Genetic Counseling; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm D (online education, pre-telephone counseling) (Experimental): Patients watch genetic testing online educational video, receive pre-telephone genetic counseling, and genetic testing online test results report.
  Interventions: Other: Educational Intervention; Other: Genetic Counseling; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Watch genetic testing online educational video
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Genetic Counseling — Receive post-telephone genetic counseling
  Arms: Arm B (online education, post telephone counseling); Arm C (online education, pre- and post-telephone counselling)
Other: Genetic Counseling — Receive pre-telephone genetic counseling
  Arms: Arm C (online education, pre- and post-telephone counselling); Arm D (online education, pre-telephone counseling)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well online genetics educational video with or without pre- and/or post-telephone genetics counseling works in assessing cancer-risk distress in patients with triple negative breast cancer. Online genetic education and telephone genetic counseling may help the doctors learn the stress a person feels about their risk of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To test the effects of online genetic education versus telephone genetic counseling on cancer-risk distress.

SECONDARY OBJECTIVES:

1. To test the effects of online genetic education versus telephone genetic counseling on testing completion rates.
2. To evaluate the role of psychological and social variables in women's reactions to genetic testing for ovarian cancer risk with variable education strategies.
3. To consider the effects of variations of genetic education/counseling on genetic knowledge, satisfaction with the decision to undergo testing, and family communication.
4. To examine the cancer screening and prevention behaviors, as well as cascade testing behaviors among patients who tested positive for a pathogenic variant.
5. To determine factors contributing to non-completion of genetic testing in subjects enrolled in a genetic testing trial.
6. To determine the impact of pre- and/or post-test genetic counseling on family communication, genetic testing concerns and screening behaviors.

OUTLINE: Patients are randomized into 1 of 4 arms.

ARM A: Patients watch genetic testing online educational video and receive genetic testing online test results report.

ARM B: Patients watch genetic testing online educational video, receive genetic testing online test results report, and post-telephone genetic counseling.

ARM C: Patients watch genetic testing online educational video, receive pre-telephone genetic counseling, genetic testing online test results report, and post-telephone genetic counseling.

ARM D: Patients watch genetic testing online educational video, receive pre-telephone genetic counseling, and genetic testing online test results report.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 or older. Note: Participants must meet each of Criteria 1-4.
* Have access to a healthcare provider and be willing to share genetic results with that provider
* Have at least one ovary
* Have a valid United States mailing address for receipt of saliva kit
* Participants must meet any one of the following 6 criteria:
* Diagnosed with breast cancer at age 45 or younger
* Diagnosed with triple negative (negative for estrogen receptor, progesterone receptor and not human epidermal growth factor receptor 2 [Her2] amplified) breast cancer at 60 or younger
* Have one blood relative with a mutation in BRCA1, BRCA2, BRIP1, PALB2, RAD51C, RAD51D, BARD1, MSH2, MSH6, MLH1, or PMS2
* Have one relative with ovarian cancer
* Have at least 2 relatives with breast cancer on the same side of the family, one of which is =< 50 years of age
* Have one male relative with breast cancer

Exclusion Criteria:

* Personal history of ovarian cancer
* Unable to read, speak, and understand English
* Unable to provide informed consent
* Unwilling to complete baseline and follow-up questionnaires
* Unable to access the internet
* Previous genetic testing or counseling regarding cancer risk
* Previous bone marrow transplant
* Previous blood transfusion (7 days prior to genetic testing)
* Active hematologic malignancy (cancer that begins in blood-forming tissue, such as leukemia or lymphoma)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Mean cancer stress scores | Up to 4 years
  Mean cancer stress scores are measured on the Impact of Events Scale (IES), a 15-item self-report measure that assesses subjective distress caused by traumatic events, which may include a positive genetic test result.There are two subscales, Intrusion and Avoidance, used to calculate a total. The range for Intrusion is 0-35 and the range for Avoidance is 0-40. The range of the total score is 0-75. Higher scores reflect more stressful impact, and therefore, a worse outcome.
  Subscales are summed to compute the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Wilke, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Swisher EM, Rayes N, Bowen D, Peterson CB, Norquist BM, Coffin T, Gavin K, Polinsky D, Crase J, Bakkum-Gamez JN, Blank SV, Munsell MF, Nebgen D, Fleming GF, Olopade OI, Law S, Zhou A, Levine DA, D'Andrea A, Lu KH. Remotely Delivered Cancer Genetic Testing in the Making Genetic Testing Accessible (MAGENTA) Trial: A Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1547-1555. doi: 10.1001/jamaoncol.2023.3748. PMID 37707822
- [Derived] Coffin T, Bowen D, Lu K, Swisher EM, Rayes N, Norquist B, Blank SV, Levine DA, Bakkum-Gamez JN, Fleming GF, I Olopade O, Romero I, D'Andrea A, Nebgen DR, Peterson C, Munsell MF, Gavin K, Crase J, Polinsky D, Lechner R. Using Social Media to Facilitate Communication About Women's Testing: Tool Validation Study. JMIR Form Res. 2022 Sep 26;6(9):e35035. doi: 10.2196/35035. PMID 36155347
- [Derived] Rayes N, Bowen DJ, Coffin T, Nebgen D, Peterson C, Munsell MF, Gavin K, Lechner R, Crase J, Polinsky D, Romero I, Blank SV, Levine DA, Norquist BM, Swisher EM, Lu KH. MAGENTA (Making Genetic testing accessible): a prospective randomized controlled trial comparing online genetic education and telephone genetic counseling for hereditary cancer genetic testing. BMC Cancer. 2019 Jul 2;19(1):648. doi: 10.1186/s12885-019-5868-x. PMID 31266460
- See also: MD Anderson Cancer Center — https://www.mdanderson.org